CLINICAL TRIAL: NCT05164107
Title: PULSE-EU - A Prospective, Non-Randomized Clinical Pilot Study to Assess Safety and Performance of a Pulsed Field Device for Global Mapping and Ablation of the Left Atrium for the Treatment of Atrial Fibrillation
Brief Title: Safety and Performance of a Pulsed Field Device for Global Mapping and Ablation of the Left Atrium for the Treatment of Atrial Fibrillation
Acronym: PULSE-EU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kardium Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DOC-140832
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
Keywords: Globe Mapping and Ablation System; Atrial Fibrillation; Pulsed Field Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Globe Mapping and Pulsed Field Ablation System (Experimental)
  Interventions: Device: Globe Mapping and Pulsed Field Ablation System (Globe PF System)

INTERVENTIONS:
Device: Globe Mapping and Pulsed Field Ablation System (Globe PF System) — During the procedure, the Globe Catheter will be delivered via standard femoral vein access and transseptal puncture. Anatomical and electrophysiological mapping of the left atrium (LA) will be followed by pulsed field ablation (PFA) to achieve pulmonary vein isolation (PVI). Additional PFA or radiofrequency (RF) ablation lesions may be created as deemed appropriate by the Investigator. Intracardiac electrogram mapping with the Globe PF System will be used to confirm PVI.

SUMMARY:
The purpose of this study is to provide clinical data pertaining to the safety and performance of the Globe Mapping and Pulsed Field Ablation System for treating subjects with atrial fibrillation (AF).

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects planned for an AF catheter ablation procedure, with a documented history of AF.

   1. Diagnosis must be confirmed within 12 months before enrollment.
   2. (Repeat ablations) Patient had 1 previous PVI procedure with cryoablation, radiofrequency ablation or pulsed field ablation
2. Subjects between 18 and 75 years of age, inclusive

Key Exclusion Criteria:

1. Patients who have contraindications to open heart surgery
2. Patients from an Intensive Care Unit
3. Patients with active systemic infection (sepsis)
4. Patients who have had previous ablation in the left or right atrium
5. Patients who are post-heart transplant or who are awaiting cardiac transplantation or other cardiac surgery
6. Patients with cardiac implants that may interfere with device delivery or positioning (e.g. atrial septal defect closure device, left atrial appendage occluder)
7. Patients with mitral valve prolapse or other heart valve abnormalities excepting mild to moderate mitral regurgitation
8. Patients with New York Heart Association Class III or IV heart failure
9. History of a documented thromboembolic event, including stroke or transient ischemic attack (TIA)
10. Bleeding disorder history
11. Patients with a known sensitivity to anesthesia or neuromuscular block agent
12. Currently undergoing long-term treatment with steroids, not including intermittent use of inhaled steroids for respiratory disease
13. Myocardial infarction within the last three months
14. Atrioventricular (AV) block II° or III°
15. Left ventricular ejection fraction (LVEF) of less than 35%
16. Unstable angina

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Rate of subjects presenting with primary safety events which are device- or procedure-related | up to 3-month visit

CONTACTS AND LOCATIONS:
Overall Officials: Motol and Homolka University Hospital, Principal Investigator — V Úvalu 84/1, 150 00 Prague 5, Czech Republic
Locations (1):
- Motol and Homolka University Hospital, Prague, Czechia